CLINICAL TRIAL: NCT03440684
Title: Effects Of The Core Stability Exercises On Balance And Hand Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ahmet GÖKKURT, Research Assistant, Gazi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Core Stability
Record Dates: First submitted 2018-02-13; First posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Healthy
Keywords: Core stability, hand, function, balance, strength
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants were included group exercise programme. The programme had been performed for 6 weeks. And participants were evaluated after exercise training programme.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy individuals (Experimental): Forty-one healthy individuals were volunteer to participate in the study and 39 of them had no neurological disease, were from 18 to 65 years old, and had no upper extremity injuries. And they have joined to exercise training during 6 weeks.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — At the beginning of the training, participants were informed about the anatomy and biomechanics of core muscles and the effectiveness core stabilization exercises.
  In all sessions, 5 minutes warm-up exercises and 5 minutes cool-down exercises were done before training. The exercises were first shown by the physiotherapist 2 to 3 repetitions and then the participants performed the exercise 10 to 12 repetitions.
  Participants were included clinical pilates exercises for 6 weeks, which would be 3 days per week. Exercise programme were managed by one and the same physiotherapist. Each week the level of difficulty of the exercises was increased according to the tolerance of the participants and new exercises were added to the program.

SUMMARY:
The core region is prescribed as a box which is formed from abdominal muscles at the front, paraspinals and glutueal muscles on the back, diaphragm on the roof, oblique abdominal muscles on sides and hip joint and pelvic girdle at the base.

With the activation of these muscles, both trunk stabilization is ensured and movement that emerges in the distal segments is supported by power generation and transfer. The location of the center of gravity in the space changes frequently with the movement of the body segments. Postural adjustments that required to restore the impaired balance due to this displacement of center of gravity, consist of lumbal stabilization with the activation of the core muscles.

The upper extremity is a body part with a wide variety of abilities. With the same basic anatomical structures, the arms, forearms, hands and fingers may function differently. The upper extremity is the primary tool that people use to manipulate the environment. Therefore, mobility comes to the forefront rather than stability in the upper extremity. On the upper extremity, the most vital component in the transition from high-level mobility to functionality is the hand. The continuity of the kinetic chain is necessary for these functions to be carried out with biomechanical and kinesiologically correct patterns.

The kinetic chain is a system that allows different body parts to produce coordinated power and collect and transfer it to the final connection point through muscle activity and body position. It is necessary to provide body stabilization by a strong core in order to achieve power transfer between the extremities and the trunk with the minimum loss of power due to this system. Core stabilization is defined as a prerequisite for the consist of movements involving the upper limb through regional biomechanical stabilization and power generation, transfer and control along the kinetic chain.

The aim of this study planned in line with the available information is to investigate the effect of core stabilization exercises applied for 6 weeks on body balance and hand functions.

DETAILED DESCRIPTION:
The core region is prescribed as a box which is formed from abdominal muscles at the front, paraspinals and glutueal muscles on the back, diaphragm on the roof, oblique abdominal muscles on sides and hip joint and pelvic girdle at the base. With the activation of these muscles, both trunk stabilization is ensured and movement that emerges in the distal segments is supported by power generation and transfer.

The location of the center of gravity in the space changes frequently with the movement of the body segments. Postural adjustments that required to restore the impaired balance due to this displacement of center of gravity, consist of lumbal stabilization with the activation of the core muscles. Kibler et al. stated that core stabilization is a key component in order to achieve balance during upper and lower limb movements and emphasized that the core is a support point for the movement of the distal segments. In addition, core stabilization exercises should be included in the balance training program as they improve body awareness and act as a muscular corset that stabilizes the body when the core area is limped or absent with limb movement.

The upper extremity is a body part with a wide variety of abilities. With the same basic anatomical structures, the arms, forearms, hands and fingers may function differently. The upper extremity is the primary tool that people use to manipulate the environment. Therefore, mobility comes to the forefront rather than stability in the upper extremity. On the upper extremity, the most vital component in the transition from high-level mobility to functionality is the hand. Daily activities such as kneading a dough, making a sculpture, cutting a meat, performing a surgical operation, thread a needle are performed manually. It also provides information about objects such as surface structures, weights, shapes, dimensions, and thermal properties. The functions of manipulating and grasping objects are functions that reveal the influence of handcraft. The continuity of the kinetic chain is necessary for these functions to be carried out with biomechanical and kinesiologically correct patterns.

The kinetic chain is a system that allows different body parts to produce coordinated power and collect and transfer it to the final connection point through muscle activity and body position. It is necessary to provide body stabilization by a strong core in order to achieve power transfer between the extremities and the trunk with the minimum loss of power due to this system. Core stabilization is defined as a prerequisite for the consist of movements involving the upper limb through regional biomechanical stabilization and power generation, transfer and control along the kinetic chain.

In a study conducted by Yuki Miyake and colleagues to investigate the effects of core stabilization exercises on upper extremity function, it was determined that only after 1 session of core stabilization training, upper-extremity functions and balance parameters have been developed in the early period. The same group of researchers underlined the lack of literature on the effects of long-term core stabilization training on balance and upper extremity functions. The aim of this study planned in line with the available information is to investigate the effect of core stabilization exercises applied for 6 weeks on body balance and hand functions.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65.

Exclusion Criteria:

* presence of neurological disease
* presence of upper extremity injury story

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2017-04-25 (Actual); Study Completion 2017-07-05 (Actual)

PRIMARY OUTCOMES:
Functional grip strength change measurement | at baseline and 6 weeks (review the change)
  Grip strength was measured by digital hand dynamometer J-Tech ™ (Midvale, USA). Participants' position was glenohumeral joint in 0° abduction and neutral rotation, elbow joint in 90° flexion, forearm and wrist in the neutral position, according to criteria determined by the American Hand Therapist Association. Three measurements were taken from dominant and non-dominant sides and the average of three measurements was recorded in kilograms.

SECONDARY OUTCOMES:
Assessment of change of static core endurance with endurance tests - 1 | at baseline and 6 weeks (review the change)
  Side Bridge Tests:
  Participants lay down on the exercise mat while their hips were 0° flexed and their knees were in full extension. Then they placed the underlying elbow joint in the flexion position so that they could support the elbow and the forearm. Participants were asked to lift their hips from the floor and to place the entire body on a flat line on their feet and elbows and to protect this position. When the participants lifted their hips from the floor, a stopwatch was started, and it was stopped when they had broken the straight position. The test was performed on the dominant and non-dominant sides. For both sides, the time in which the position was preserved was recorded as the score in seconds.
Assessment of change of static core endurance with endurance tests - 2 | at baseline and 6 weeks (review the change)
  Trunk Flexion Test:
  Participants were asked to place their knees and hips on the exercise cradle in a 90° flexion and arms crossed on the opposite shoulders. While maintaining this position, the therapist supported the upper body so as to make a 60° angle to the floor. When the support applied to the trunk was cut off, they were said to stay still at a 60˚ angle between the ground and the trunk. When the support applied to the trunk was cut off, the stopwatch was started. The stopwatch was stopped when the position deteriorated, and the elapsed time was recorded in seconds.
Assessment of change of static core endurance with endurance tests - 3 | at baseline and 6 weeks (review the change)
  Trunk Extension Test (Biering-Sorensen Test) Participants lay on face on the test bed in a position which their knee and hip joints were in full extension and their ankles, knees, hips and the upper-part of iliac crest were about to touch the test bed. The upper bodies were placed in a resting position on a stool placed in front of the test bed. Later, participants were asked to position their arms in the opposite T position and stay still in this position by bringing their bodies to the horizontal line. When the line occurred, a stopwatch was started, and it was stopped when the position was disturbed. The score was recorded in seconds.
Assessment of change of static core endurance with endurance tests - 4 | at baseline and 6 weeks (review the change)
  Prone Bridge Test Participants were supported by their elbows and extended to the exercise mat in the prone position. The amount of openness of the elbows was determined as the shoulder width. Participants were asked to remove their hips from the ground and form a linear line when their forearms and toes were in contact with the ground. When the linear line was formed, the stopwatch was started and stopped when the positions were broken. The position protection duration was recorded as the score in seconds.
Assessment of change of dynamic core endurance with endurance tests | at baseline and 6 weeks (review the change)
  Modified Push-Ups Test Participants cross over their legs while the knees are flexed on the exercise mat and stretch out in a prone position. Then participants were asked to put their hands around and to lift their heads, trunk and hips in such a way so as to create a straight line by extending their elbows. The number of repetitions made within thirty seconds was recorded as the result.
  Sit-Ups Test Participants stretched over the supine position so that the knees on the exercise mat would be 90° flexed. They were asked to place their hands next to their heads and to perform body flexing when the therapist was supporting their feet. The number of repetitions made within thirty seconds was recorded as the result.
Assessment of balance change | at baseline and 6 weeks (review the change)
  Biodex ™ Biosway ™ (Shirley, USA) was used for balance evaluation in our study. Only postural sway of the participants was evaluated within the scope of the study. During the postural sway evaluation, the amount of displacement of the center of gravity is automatically calculated by the device.
  The aim of the balance assessment in this study was to evaluate the postural sway during hand function. Thus, the participant performed PPT that placed on a 70-cm height table in front of participant while standing on the platform. The measurement time of postural sway was set to 30 seconds according to the PPT application period and the measurement was repeated twice. Between the two assessments, participants were given a rest period of 10 seconds. After the evaluation, three different scores were created by the device, anteroposterior, mediolateral and overall. The scores obtained were recorded.
Functional hand ability change assessment - 1 | at baseline and 6 weeks (review the change)
  Nine Hole Peg Test (NHPT) and Purdue Pegboard Test (PPT), which are speed dependent hand function tests, were used to evaluate the functional ability of the hand. NHPT is a test with 9 holes and 9 pins. While participants are sitting in the chair, they pull the pins out of the holes in the fastest way on the table and then push them back into the holes. The first evaluation was called an experiment and the test duration was not calculated. At the second evaluation, chronometer started when the participant touched the first pine, and it stopped when the last pine was placed. Scores were recorded as the time in seconds. The test was performed for the dominant and non-dominant sides.
Functional hand ability change assessment - 2 | at baseline and 6 weeks (review the change)
  Another performance test is PPT which consists of pins, pulls and cap nuts and can make 4 different evaluations. In this study, only one of the subtests was used without using pulls and cap nuts. How many of 40 pins were inserted to 40 holes within 30 secs by participants was counted. The test was performed on a 70-cm high table placed in front of the participant in the standing position during the balance assessment [16]. The evaluation was only performed in dominant side and was repeated 2 times. The result score was calculated by taking the average of the number of pins the participant can put in 30 seconds in 2 measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi Üniversitesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Participants' information collected for this study. It's not planned that share or use this information by investigators.

REFERENCES:
- [Background] Akuthota V, Ferreiro A, Moore T, Fredericson M. Core stability exercise principles. Curr Sports Med Rep. 2008 Feb;7(1):39-44. doi: 10.1097/01.CSMR.0000308663.13278.69. PMID 18296944
- [Background] Kibler WB, Press J, Sciascia A. The role of core stability in athletic function. Sports Med. 2006;36(3):189-98. doi: 10.2165/00007256-200636030-00001. PMID 16526831
- [Background] Shinkle J, Nesser TW, Demchak TJ, McMannus DM. Effect of core strength on the measure of power in the extremities. J Strength Cond Res. 2012 Feb;26(2):373-80. doi: 10.1519/JSC.0b013e31822600e5. PMID 22228111
- [Background] Miyake Y, Kobayashi R, Kelepecz D, Nakajima M. Core exercises elevate trunk stability to facilitate skilled motor behavior of the upper extremities. J Bodyw Mov Ther. 2013 Apr;17(2):259-65. doi: 10.1016/j.jbmt.2012.06.003. Epub 2012 Jul 10. PMID 23561876
- [Background] McGill SM, Childs A, Liebenson C. Endurance times for low back stabilization exercises: clinical targets for testing and training from a normal database. Arch Phys Med Rehabil. 1999 Aug;80(8):941-4. doi: 10.1016/s0003-9993(99)90087-4. PMID 10453772
- [Background] Biering-Sorensen F. Physical measurements as risk indicators for low-back trouble over a one-year period. Spine (Phila Pa 1976). 1984 Mar;9(2):106-19. doi: 10.1097/00007632-198403000-00002. PMID 6233709
- [Background] Bliss LS, Teeple P. Core stability: the centerpiece of any training program. Curr Sports Med Rep. 2005 Jun;4(3):179-83. doi: 10.1007/s11932-005-0064-y. PMID 15907272
- [Background] Hodges PW, Richardson CA. Feedforward contraction of transversus abdominis is not influenced by the direction of arm movement. Exp Brain Res. 1997 Apr;114(2):362-70. doi: 10.1007/pl00005644. PMID 9166925
- [Background] TIFFIN J, ASHER EJ. The Purdue pegboard; norms and studies of reliability and validity. J Appl Psychol. 1948 Jun;32(3):234-47. doi: 10.1037/h0061266. No abstract available. PMID 18867059
- See also: Owsley, A. (2005). An introduction to clinical Pilates. Athletic Therapy Today. 10(4): p. 19-25. — https://doi.org/10.1123/att.10.4.19